CLINICAL TRIAL: NCT00671203
Title: Prevention of Colon Ischemia During Aortic Aneurysm (AAA) Repair
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectros Corporation (Industry)
Collaborators: Stanford University (Other); University of California (Other)
Responsible Party: Spectros Corporation, Clinical Studies Director
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAA-002; NIH DK068927
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Colon Ischemia; Aortic Aneurysm
Keywords: Tissue oximetry; Ischemia; Aortic Aneurysm Repair; Aortic Stent; Vascular Stent; Aortic graft; Vascular graft
MeSH Terms: conditions — Aortic Aneurysm; Ischemia | interventions — Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Reestablish colon blood flow — If ischemia is detected, and the detection in consistent with the physician's clinical view, blood flow to the colon is established using any of the known techniques that would be used had the diagnosis been made in the absence of T-Stat, which include changes in the deployment of stents and/or coils, reanastomosis, reimplantation, or stenting, of obstructed vessels, or other established techniques.
  Other Names: T-Stat Ischemia Detection System (#303); T-Stat 5mm sensor catheter (#CTH-060)

SUMMARY:
Patients undergoing surgery on their Aorta can get ischemia, a lack of blood flow, to their intestines and colon. This is very serious, as 2 out of 3 patients who have this problem die before leaving the hospital. A device developed by Spectros, called T-Stat, is approved by the US FDA to detect ischemia, and has been reported to detect ischemia in AAA aneurysm surgery and stenting, allowing the surgeon or interventional radiologist to take action quickly, while the colon ischemia is still treatable.

This purpose of this study is to establish how T-Stat can best be used to prevent deaths.

ELIGIBILITY:
Inclusion Criteria:

* Aortic Aneurysm, intact or ruptured
* Repair by catheter based stent or by open surgery during monitoring
* Patent rectum
* Absence of rectal bleeding

Exclusion Criteria:

* Lack of informed consent
* Rectal bleeding
* Obstructed rectum

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Detect colon ischemia early | Just before, and during, surgery or stenting

SECONDARY OUTCOMES:
Allows change in the untreated course of colon ischemia | 28 days or discharge from hospital

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California at Davis Medical Center, Davis, California
  - Stanford University Vascular Surgery, Palo Alto, California

REFERENCES:
- [Background] Friedland S, Benaron D, Coogan S, Sze DY, Soetikno R. Diagnosis of chronic mesenteric ischemia by visible light spectroscopy during endoscopy. Gastrointest Endosc. 2007 Feb;65(2):294-300. doi: 10.1016/j.gie.2006.05.007. Epub 2006 Sep 20. PMID 17137857
- [Background] Benaron DA, Parachikov IH, Friedland S, Soetikno R, Brock-Utne J, van der Starre PJ, Nezhat C, Terris MK, Maxim PG, Carson JJ, Razavi MK, Gladstone HB, Fincher EF, Hsu CP, Clark FL, Cheong WF, Duckworth JL, Stevenson DK. Continuous, noninvasive, and localized microvascular tissue oximetry using visible light spectroscopy. Anesthesiology. 2004 Jun;100(6):1469-75. doi: 10.1097/00000542-200406000-00019. PMID 15166566
- [Result] Lee ES, Bass A, Arko FR, Heikkinen M, Harris EJ, Zarins CK, van der Starre P, Olcott C. Intraoperative colon mucosal oxygen saturation during aortic surgery. J Surg Res. 2006 Nov;136(1):19-24. doi: 10.1016/j.jss.2006.05.014. Epub 2006 Sep 15. PMID 16978651
- [Result] Lee ES, Pevec WC, Link DP, Dawson DL. Use of T-Stat to predict colonic ischemia during and after endovascular aneurysm repair: a case report. J Vasc Surg. 2008 Mar;47(3):632-4. doi: 10.1016/j.jvs.2007.09.037. PMID 18295116
- See also: Spectros Corporation T-Stat Web Site — http://www.spectros.com